CLINICAL TRIAL: NCT06339294
Title: Efficacy of Pyodine Soaked Gelfoam vs Single Topical Application of Clotrimazole in Treatment of Otomycosis: a Randomized Controlled Clinical Trial
Brief Title: Efficacy of Pyodine Soaked Gelfoam vs Single Topical Application of Clotrimazole in Otomycosis Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rawalpindi Medical College (Other)
Responsible Party: Principal Investigator, Dr Zuneera Shabbir, Primary Investigator, Rawalpindi Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZShabbir
Record Dates: First submitted 2024-03-17; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Otomycosis
Keywords: Otomycosis; clotrimazole ointment; povidone iodine
MeSH Terms: conditions — Otomycosis | interventions — Povidone-Iodine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (clotrimazole ointment group) (Experimental): Clotrimzole ointment
  1ml dose Frequency one time application Duration one time application with aural toilet after 7 days
  Interventions: Drug: Clotrimazole Cream
- Group B(Povidone Iodine group) (Experimental): Povidone iodine solution
  1ml dose Frequency one time application Duration one time application with aural toilet after 7 days
  Interventions: Drug: Povidone-Iodine

INTERVENTIONS:
Drug: Clotrimazole Cream — Single time application of clotrimazole ointment was done after aural toilet in external auditory canal via IV catheter
  Arms: Group A (clotrimazole ointment group)
Drug: Povidone-Iodine — Gelfoam soaked pyodine solution was placed in external auditory canal after aural toilet
  Arms: Group B(Povidone Iodine group)

SUMMARY:
Background and Objectives To compare the efficacy of gel foam-soaked pyodine with a single topical application of clotrimazole ointment.

Subjects and Methods This randomized controlled trial will include 90 patients presenting to ENT OPD with complaints of earache, watery ear discharge, pruritis, and ear blockage and will be clinically diagnosed as a case of otomycosis on otoscopy. The external auditory canal of the patient will be cleared of fungal debris via suction before treatment In Group A ear canal will be filled with 1% clotrimazole ointment by using an IV catheter and syringe and in Group B pyodine-soaked gel foam will be placed in the external auditory canal. The patients will be followed up on post-treatment days 7 and 14.

DETAILED DESCRIPTION:
INTRODUCTION:

Otomycosis, external auditory canal fungal infection is a recurrent and prevalent condition affecting 9%to 27.2% of patients worldwide. Use of topical antibiotics, humid conditions, and trauma to the external auditory canal are well-recognized risk factors for this disease. Aspergillus nigar (60-90%), and Candida species (10-40%) are the most commonly isolated pathogens in patients with otomycosis. Otomycosis presents with bothersome symptoms such as pruritis, watery ear discharge, otalgia, and ear blockage which significantly impairs the patient's quality of life Therapeutic approaches for fungal ear infections include aural toilet, withholding topical antibiotics, starting topical antifungals, and enhancing patient well-being and cleanliness Multiple treatment options are available for the treatment of otomycosis but the recurrence rate of the disease is high. While several antifungal agents have been employed for its treatment, due to a lack of efficacy comparison it is difficult to select an appropriate option The choice of therapy plays an important role in achieving rapid symptom resolution and complete fungal eradication. Clotrimazole, a conventional antifungal agent, has been widely employed, but its efficacy is not always optimal. For topical treatment compliance of the patient and proper application of medication is also an important factor affecting the efficacy of the drug. Conversely, the utilization of pyodine-soaked Gelfoam is a novel approach that offers several advantages, including sustained drug release better drug penetration, and decreased risk of resistance as in the case of antifungals.

Due to reduced compliance of the patients and ineffective technique of using topical antifungal otomycosis has a high rate of treatment failure and recurrence. Topical clotrimazole drops and povidine iodine solution have been compared for their efficacy in the past but a single topical application has not been compared until now. In this pursuit, we present a rigorous and comprehensive clinical trial designed to evaluate the comparative efficacy of two distinct treatment modalities: pyodine-soaked Gelfoam and a single topical application of 1% clotrimazole. The rationale behind this study is to address the escalating concerns regarding treatment-resistant otomycosis, as well as the need for cost-effective and practical solutions By addressing the question of which treatment is superior, this study endeavors to optimize the management of otomycosis, ensuring better patient outcomes and reduced healthcare costs.

MATERIAL & METHODS:

The main objective of this study is to evaluate the effectiveness of povidone iodine-soaked gel foam vs clotrimazole ointment in the management of otomycosis. A randomized controlled study was done in the ENT Department of Benazir Bhutto Hospital Rawalpindi over a period of 6 months from June 2023 to December 2023.

Individuals with a clinical otomycosis diagnosis were recruited for the study. Individuals with active CSOM, external auditory canal abnormalities, and hearing aids were excluded from the study. A sample size of 90 patients was calculated. After approval from the ethical review board, patients were selected from the ENT clinic of Benazir Bhutto Hospital and enrolled in two treatment groups after obtaining informed consent. Complete history was taken from the patients and the ear canal was assessed by otoscopy. The aural toilet of all patients was done via suctioning of the ear canal. In Group A patient's ear canal was filled with 1% clotrimazole ointment by using an Intravenous catheter and syringe In Group B pyodine solution-soaked gel foam was placed in the external auditory canal. Followup of patients was done on the 7th and 14th post-treatment days otoscopy was performed and post-treatment symptom resolution and ear canal condition were assessed. Patients were allocated to three groups based on their clinical outcomes

Good response Patients with a dry EAC and tympanic membrane intact

Partial Response:

Patients with scanty discharge but not completely dry EAC

No Response:

Patients with unusually high EAC Exudation

ELIGIBILITY:
Inclusion Criteria:

* All patients with clinical diagnosis of otomycosis via otoscopy

Exclusion Criteria:

* Active CSOM
* External auditory canal abnormalities
* Patients on hearing aids

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Treatment Response Based on Otoscopy | 7th and 14th post treatment day
  Good response Patients with a dry EAC and tympanic membrane intact with no fungal spores
  Partial Response:
  Patients with scanty discharge but not completely dry EAC with no fungal spores
  No Response:
  Patients with unusually high EAC Exudation with fungal spores present

SECONDARY OUTCOMES:
Condition of External Auditory Canal | 7th and 14th post treatment day
  Condition of External Auditory canal will be assessed via otoscop External auditory canal edema and erythema: Present or not Tympanic membrane congestion: Present or not Purulent discharge: Present or Not

CONTACTS AND LOCATIONS:
Overall Officials: Zuneera Shabbir PGR, MBBS, Principal Investigator — Rawalpindi Medical College
Locations (1):
- Benazir Bhutto Hospital, Rawalpindi, Punjab/46000, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jwery AK. Various topical antifungal agents in otomycosis, which is the best? J Pak Med Assoc. 2021 Dec;71(Suppl 8)(12):S32-S34. PMID 35130214
- [Background] Haq M, Deshmukh P. Review of Recurrent Otomycosis and Clotrimazole in Its Treatment. Cureus. 2022 Oct 9;14(10):e30098. doi: 10.7759/cureus.30098. eCollection 2022 Oct. PMID 36381881
- [Result] Chavan RP, Ingole SM, Kanchewad Resident GS. Single Topical Application of 1% Clotrimazole Cream in Otomycosis. Indian J Otolaryngol Head Neck Surg. 2023 Apr;75(Suppl 1):147-154. doi: 10.1007/s12070-022-03206-x. Epub 2022 Dec 8. PMID 36532230

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/94/NCT06339294/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-16): https://cdn.clinicaltrials.gov/large-docs/94/NCT06339294/ICF_001.pdf